CLINICAL TRIAL: NCT05354453
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 1839100 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 1839100 Are Tolerated (1490-0001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1490-0001; 2021-006294-27 (EudraCT Number)
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Healthy
MeSH Terms: interventions — allyl isothiocyanate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SRD Part (Experimental): Single-rising dose (SRD)
  Interventions: Drug: BI 1839100
- SRD Part: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Skin Challenge Part (Experimental)
  Interventions: Drug: BI 1839100; Drug: allyl isothiocyanate (AITC)
- Skin Challenge Part: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: allyl isothiocyanate (AITC)

INTERVENTIONS:
Drug: BI 1839100 — BI 1839100
  Arms: SRD Part; Skin Challenge Part
Drug: Placebo — Placebo
  Arms: SRD Part: Placebo; Skin Challenge Part: Placebo
Drug: allyl isothiocyanate (AITC) — allyl isothiocyanate (AITC)
  Arms: Skin Challenge Part; Skin Challenge Part: Placebo

SUMMARY:
This trial starts the clinical development of BI 1839100. Effects of single rising doses of BI 1389100 on safety, tolerability and pharmacokinetics will be assessed as basis for further development in patients with pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 31.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male subjects who meet any of the following criteria for a highly effective contraception from the first administration of trial medication until 90 days after trial completion:

  * Willing to use a medically accepted method of contraception. Acceptable methods of contraception for use by male subjects include sexual abstinence, a vasectomy performed at least 1 year prior to dosing, and barrier contraception (condom)
  * Subjects who are not vasectomised or sexually abstinent have to ensure that an additional acceptable method of contraception (in addition to male condom) will be used by his female partner such as intrauterine device (IUD), surgical sterilisation (including hysterectomy), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 month prior to drug administration or postmenopausal status of female partner (defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm (subjects with heart rate values between 45 and 50 bpm may only be enrolled in case they have a normal thyroid function, no clinical symptoms associated with the bradycardia and no apparent signs of other diseases causing bradycardia such as hypothyroidism or heart conduction abnormalities)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 10 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 1839100 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 4 days
Maximum measured concentration of BI 1839100 in plasma (Cmax) | up to 4 days
Time from dosing to maximum measured concentration of BI 1839100 in plasma (tmax) | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com